CLINICAL TRIAL: NCT00887536
Title: A Phase III Clinical Trial Comparing the Combination of TC Plus Bevacizumab to TC Alone and to TAC for Women With Node-Positive or High-Risk Node-Negative, HER2-Negative Breast Cancer
Brief Title: A Clinical Trial Comparing the Combination of TC Plus Bevacizumab to TC Alone and to TAC for Women With Node-Positive or High-Risk Node-Negative, HER2-Negative Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Genentech, Inc. (Industry); US Oncology Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP B-46-I; USOR 07132
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: National Surgical Adjuvant Breast and Bowel Project (NSABP); Taxotere; Docetaxel; Doxorubicin; Cyclophosphamide; Bevacizumab; Breast Neoplasms; Adenocarcinoma; Breast Diseases; Carcinoma; HER2 negative; Node negative; High risk node positive; Adjuvant Therapy
MeSH Terms: conditions — Breast Neoplasms; Adenocarcinoma; Breast Diseases; Carcinoma | interventions — Bevacizumab; Docetaxel; Doxorubicin; Cyclophosphamide; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: TAC then pegfilgrastim (Active Comparator): docetaxel, doxorubicin, cyclophosphamide, and pegfilgrastim/filgrastim
  Interventions: Drug: docetaxel; Drug: doxorubicin; Drug: cyclophosphamide; Drug: pegfilgrastim
- Group 2: TC (Active Comparator): docetaxel and cyclophosphamide
  Interventions: Drug: docetaxel; Drug: cyclophosphamide
- Group 3: TC + bevacizumab (Experimental): docetaxel, cyclophosphamide, and bevacizumab
  Interventions: Drug: bevacizumab; Drug: docetaxel; Drug: cyclophosphamide

INTERVENTIONS:
Drug: bevacizumab — bevacizumab 15 mg/kg IV every 21 days for 6 cycles followed by bevacizumab 15 mg/kg IV every 21 days until 1 year following the first dose of bevacizumab
  Arms: Group 3: TC + bevacizumab
Drug: docetaxel — docetaxel 75 mg/m2 IV every 21 days for 6 cycles
  Other Names: T
Drug: doxorubicin — doxorubicin 50 mg/m2 IV every 21 days for 6 cycles
  Other Names: A
  Arms: Group 1: TAC then pegfilgrastim
Drug: cyclophosphamide — Group 1: cyclophosphamide 500 mg/m2 IV every 21 days for 6 cycles
  Group 2 and 3: cyclophosphamide 600 mg/m2 IV every 21 days for 6 cycles
  Other Names: C
Drug: pegfilgrastim — pegfilgrastim 6 mg subcutaneous (SC) Day 2 every 21 days for 6 cycles [filgrastim (Neupogen®) 5 mcg/kg Days 2-10 may be given in lieu of pegfilgrastim (Neulasta®), but pegfilgrastim is preferred.]
  Arms: Group 1: TAC then pegfilgrastim

SUMMARY:
The main purpose of this study is to learn if adding bevacizumab to standard treatment with chemotherapy (docetaxel, doxorubicin, and cyclophosphamide) for early stage HER2-negative breast cancer will prevent breast cancer from returning. A second purpose of this study is to learn if adding bevacizumab to treatment with chemotherapy will help women with HER2-negative breast cancer live longer. The researchers also want to learn about the side effects of the combination of drugs used in this study.

DETAILED DESCRIPTION:
The B-46-I/07132 study, a multicenter, open-label, randomized Phase III, adjuvant therapy trial, will compare the value of adding bevacizumab to a non-anthracycline-based chemotherapy regimen relative to the same chemotherapy without bevacizumab and relative to an anthracycline-based chemotherapy regimen in women with resected node-positive or high-risk node-negative, HER2-negative breast cancer. This trial will determine whether the addition of bevacizumab to a regimen of docetaxel and cyclophosphamide (TCB) improves invasive disease-free survival relative to docetaxel and cyclophosphamide alone (TC). A secondary aim will be to determine whether the addition of bevacizumab to TC improves invasive disease-free survival compared to a regimen of docetaxel, doxorubicin, and cyclophosphamide (TAC). Other secondary aims include whether TCB improves disease-free survival, overall survival, and recurrence-free interval relative to TC alone and to TAC. The toxicities of the three regimens will also be compared.

Patients in the B-46-I/07132 study will be randomized to one of three treatment regimens: Group 1 patients will receive 6 cycles of TAC administered every 21 days (docetaxel 75 mg/m2, doxorubicin 50 mg/m2, and cyclophosphamide 500 mg/m2); Group 2 patients will receive 6 cycles of TC administered every 21 days (docetaxel 75 mg/m2, cyclophosphamide 600 mg/m2); and Group 3 patients will receive 6 cycles of TCB every 21 days with bevacizumab therapy continuing every 21 days after completion of chemotherapy until 1 year following the first dose (docetaxel 75 mg/m2, cyclophosphamide 600 mg/m2, and bevacizumab 15 mg/kg). Primary prophylaxis with pegfilgrastim or filgrastim is required for Group 1 patients (optional for patients in Groups 2 and 3). Patients will also receive adjuvant radiation therapy as clinically indicated and endocrine therapy for hormone receptor-positive tumors.

Tumor samples will be submitted for correlative science studies to evaluate predictors of study therapy benefit. Submission of a tumor sample is a study requirement for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be female.
* The patient must be greater than or equal to 18 years of age and less than or equal to 70 years of age.
* The patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* The tumor must be unilateral invasive adenocarcinoma of the breast on histologic examination.
* The breast cancer must be HER2-negative based on current American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) Guideline Recommendations for Human Epidermal Growth Factor Receptor 2 Testing in Breast Cancer. If the result of the in situ hybridization testing (FISH, chromagen in situ hybridization (CISH), or other) is equivocal, the patient is eligible if there is no plan to administer HER2-targeted therapy.
* All of the following staging criteria (according to the 6th edition of the American Joint Committee on Cancer (AJCC) Cancer Staging Manual) must be met: By pathologic evaluation, primary tumor must be pT1-3; By pathologic evaluation, ipsilateral nodes must be pN0, pN1 (pN1mi, pN1a, pN1b, pN1c), pN2a, pN3a, or pN3b. If pN0, at least one of the following criteria must be met: ER negative and PgR negative; or Pathologic tumor size greater than 2.0 cm; or T1c (pathologic tumor size greater than 1.0 cm but less than or equal to 2.0 cm) and ER positive (PgR status may be positive or negative) and either Oncotype DX® Recurrence Score of greater than or equal to 25 or grade 3 histology.
* Patients must have undergone either a total mastectomy or breast-conserving surgery (lumpectomy).
* For patients who undergo lumpectomy, the margins of the resected specimen must be histologically free of invasive tumor and DCIS as determined by the local pathologist. If pathologic examination demonstrates tumor at the line of resection, additional operative procedures must be performed to obtain clear margins. If tumor is still present at the resected margin after re-excision(s), the patient must undergo total mastectomy to be eligible. (Patients with margins positive for lobular carcinoma in situ [LCIS] are eligible without additional resection.)
* For patients who undergo mastectomy, margins must be histologically free of invasive tumor and DCIS.
* Patients must have completed one of the following procedures for evaluation of pathologic nodal status: Sentinel lymphadenectomy alone if pathologic nodal staging based on sentinel lymphadenectomy is pN0, pN1mi, or pN1b; Sentinel lymphadenectomy followed by removal of additional non-sentinel lymph nodes if the sentinel node (SN) is positive; or Axillary lymphadenectomy without SN isolation procedure.
* The interval between the last surgery for breast cancer (treatment or staging) and randomization must be at least 28 days but no more than 84 days.
* Patients must have ER analysis performed on the primary tumor prior to randomization. If ER analysis is negative, then PgR analysis must also be performed. (Either a core biopsy or surgical resection specimen can be used for ER/PgR testing.)
* The most recent postoperative blood counts must meet the following criteria: Absolute neutrophil count (ANC) must be greater than or equal to 1200/mm3; platelet count must be greater than or equal to 100,000/mm3; and hemoglobin must be greater than or equal to 10 g/dL.
* The following criteria for evidence of adequate hepatic function must be met based on the results of the most recent postoperative tests: total bilirubin must be less than or equal to upper limits of normal (ULN)for the lab unless the patient has a bilirubin elevation less than ULN to 1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and alkaline phosphatase must be less than or equal to 2.5 x ULN for the lab; and AST must be less than or equal to 1.5 x ULN for the lab. Alkaline phosphatase and aspartate transaminase (AST) may not both be greater than the ULN. For example, if the alkaline phosphatase is greater than the ULN but less than or equal to 2.5 x ULN, then the AST must be less than or equal to the ULN. If the AST is greater than the ULN but less than or equal to 1.5 x ULN, then the alkaline phosphatase must be less than or equal to ULN.
* Patients with AST or alkaline phosphatase greater than ULN are eligible for inclusion in the study if liver imaging (CT, MRI, PET-CT, or PET scan) does not demonstrate metastatic disease and the requirements for adequate hepatic function are met.
* Patients with alkaline phosphatase that is greater than ULN but less than or equal to 2.5 x ULN are eligible for inclusion in the study if a bone scan, PET-CT, or PET scan does not demonstrate metastatic disease.
* The most recent postoperative serum creatinine must be less than or equal to ULN for the lab.
* A urine sample must be tested for proteinuria by the dipstick method. Eligibility must be based on the most recent postoperative test result(s) performed within 6 weeks prior to randomization. Urine dipstick must indicate 0-1+ protein. If dipstick reading is greater than or equal to 2+, a 24-hour urine specimen must be collected and must demonstrate less than 1 gram of protein.
* Left ventricular ejection fraction (LVEF) assessment by 2-D echocardiogram or multigated acquisition (MUGA) scan must be performed within 90 days prior to randomization. The LVEF must be greater than or equal to 50% regardless of the facility's lower limits of normal (LLN).

Exclusion Criteria:

* T4 tumors including inflammatory breast cancer.
* Definitive clinical or radiologic evidence of metastatic disease.
* Synchronous or metachronous contralateral invasive breast cancer. (Patients with synchronous and/or metachronous contralateral DCIS are eligible.)
* Any history of ipsilateral invasive breast cancer or ipsilateral DCIS.
* History of non-breast malignancies within 5 years prior to randomization, except for the following: carcinoma in situ of the cervix, colorectal carcinoma in situ, melanoma in situ, and basal cell and squamous cell carcinomas of the skin.
* Previous therapy with anthracyclines, taxanes, or bevacizumab for any malignancy.
* Chemotherapy administered for the currently diagnosed breast cancer prior to randomization.
* Continued therapy with any hormonal agent such as raloxifene or tamoxifen (or other SERM) or an aromatase inhibitor. (Patients are eligible if these medications are discontinued prior to randomization.)
* Any sex hormonal therapy, e.g., birth control pills, ovarian hormone replacement therapy. Patients are eligible if these medications are discontinued prior to randomization.
* Active hepatitis B or hepatitis C with abnormal liver function tests.
* Cardiac disease (history of and/or active disease) that would preclude the use of the drugs included in the treatment regimens. This includes but is not confined to 1) Active cardiac disease: angina pectoris that requires the use of anti-anginal medication; ventricular arrhythmias except for benign premature ventricular contractions; supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication; conduction abnormality requiring a pacemaker; valvular disease with documented compromise in cardiac function; and symptomatic pericarditis, 2) History of cardiac disease: myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of left ventricular (LV) function; history of documented congestive heart failure (CHF); and documented cardiomyopathy.
* Uncontrolled hypertension defined as systolic BP greater than 150 mmHg or diastolic BP greater than 90 mmHg, with or without anti-hypertensive medication. Patients with initial BP elevations are eligible if initiation or adjustment of BP medication lowers pressure to meet entry criteria.
* History of hypertensive crisis or hypertensive encephalopathy.
* History of transient ischemic attack (TIA) or cerebrovascular accident (CVA).
* History of any arterial thrombotic event within 12 months prior to randomization.
* Symptomatic peripheral vascular disease.
* Intrinsic lung disease resulting in dyspnea.
* Unstable diabetes mellitus.
* Active infection or chronic infection requiring suppressive antibiotics.
* History of a major organ allograft or condition requiring chronic immunosuppression, e.g., kidney, liver, lung, heart, bone marrow transplant, or autoimmune diseases. (Patients who have received corneal transplants, cadaver skin, or bone transplants are eligible.)
* Any significant bleeding within 180 days prior to randomization, exclusive of menorrhagia in premenopausal women.
* Non-healing wound, skin ulcers, or incompletely healed bone fracture.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to the planned start of study therapy.
* Anticipation of need for major surgical procedures during study therapy and for at least 3 months following completion of bevacizumab.
* Gastroduodenal ulcer(s) documented by endoscopy to be active within 6 months before randomization.
* History of GI perforation, abdominal fistulae, or intra-abdominal abscess.
* Known bleeding diathesis or coagulopathy.
* Requirement for therapeutic doses of coumadin or equivalent.
* Sensory/motor neuropathy greater than or equal to grade 2, as defined by the NCI Common Terminology Criteria for Adverse Events (CTCAE) v3.0.
* Conditions that would prohibit administration of corticosteroids.
* Chronic daily treatment with corticosteroids (dose of greater than or equal to 10 mg/day methylprednisolone equivalent) (excluding inhaled steroids).
* History of hypersensitivity reaction to drugs formulated with polysorbate 80.
* Pregnancy or lactation at the time of study entry.
* Other non-malignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow-up.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.
* Use of any investigational product within 4 weeks prior to randomization.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1613 (Actual)
Dates: Start 2009-05; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Invasive disease-free survival(IDFS)relative to the TAC chemotherapy regimen alone | Every 12 months until recurrence

SECONDARY OUTCOMES:
Invasive disease-free survival (IDFS) relative to the TAC chemotherapy regimen | Every 12 months until recurrence
Disease-free survival (DFS-DCIS) relative to the TC alone regimen | Every 12 months until recurrence
Overall survival (OS) relative to the TC alone regimen | Every 12 months from randomization until death from any cause
OS relative to the TAC regimen | Every 12 months from randomization until death from any cause
Recurrence-free interval (RFI) relative to the TC alone regimen | Every 12 months, from randomization to local, regional, or distant recurrence
RFI relative to the TAC regimen | Every 12 months, from randomization to local, regional, or distant recurrence
Develop molecular predictive markers for the degree of benefit from TCB over TC or TAC | 6 years
Provide the efficacy data from Group 1 patients and Group 2 patients enrolled in B-46-I/07132 to US Oncology Research, Inc. (USOR) for a planned combined analysis with efficacy data from patients receiving the same regimens in the USOR 06-090 trial | 10 years
Toxicity associated with each of the regimens | Every 6 months
Determine the role of topoisomerase II alpha (TOP2A) in prognosis and prediction of degree of benefit from TAC over TC | 6 years
Develop predictive markers for benefit from doxorubicin | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (531):
- United States (520):
  - Birmingham Hematology and Oncology, Bessemer, Alabama
  - Birmingham Hematology and Oncology, Birmingham, Alabama
  - Birmingham Hematology and Oncology - Brookwood, Birmingham, Alabama
  - Birmingham Hematology and Oncology - Princeton, Birmingham, Alabama
  - Birmingham Hematology and Oncology - Montclair, Birmingham, Alabama
  - Birmingham Hematology and Oncology - Pilot, Birmingham, Alabama
  - Clearview Cancer Institute- Huntsville, Huntsville, Alabama
  - Northern Arizona Hematology & Onclogy Associates, Flagstaff, Arizona
  - Arizona Oncolocy (CASA-Green Valley), Green Valley, Arizona
  - Arizona Oncology (CASA- Oro Valley), Oro Valley, Arizona
  - Hematology Oncology Associates, Phoenix, Arizona
  - Northern Arizona Hematology & Oncology Associates, Prescott Valley, Arizona
  - Arizona Oncology (CASA-Safford), Safford, Arizona
  - Hematology Oncology Associates, Scottsdale, Arizona
  - Northern Arizona Hematology & Oncology Associates, Sedona, Arizona
  - Arizona Oncology Associates - Rudasill, Tucson, Arizona
  - Arizona Oncology Associates - Carondelet, Tucson, Arizona
  - Arizona Oncology (CASA-Craycroft), Tucson, Arizona
  - Arizona Oncology (CASA-Office Only), Tucson, Arizona
  - Arizona Oncology - CASA St. Mary's, Tucson, Arizona
  - Central Hematology/Oncology Medical Group, Inc., Alhambra, California
  - Kaiser Permanente Deer Valley Med Center, Antioch, California
  - Comp Blook and Cancer Center, Bakersfield, California
  - Southwest Cancer Care (E. Grand), Escondido, California
  - Kaiser Permanente Fremont, Fremont, California
  - St. Jude Heritage Healthcare, Fullerton, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Pacific Shores Medical Group, Huntington Beach, California
  - Southern California Permanente Medical Group, Irvine, California
  - Wilshire Oncology Medical Group (Business Office), La Verne, California
  - Antelope Valley Cancer Center, Lancaster, California
  - Breastlink Medical Group, Incorporated at Long Beach Memorial Medical Center, Long Beach, California
  - Todd Cancer Institute at Long Beach Memorial Med Cent, Long Beach, California
  - Pacific Shores Medical Group, Long Beach, California
  - Pacific Shores Medical Group, Los Alamitos, California
  - TORI- N Valley Hematology Oncology Med Group, Mission Hills, California
  - TORI - Oncology Care Medical Assoc., Montebello, California
  - Southwest Cancer Care (Medical Center), Murrieta, California
  - NValley Hematology/Oncology Medical Group, Northridge, California
  - Kaiser Permanente-Oakland, Oakland, California
  - St. Joseph Hospital, Orange, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Stanford University Medical Center, Palo Alto, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Roseville, Roseville, California
  - Sutter Medical Center, Sacramento, California
  - Kaiser Permanente, South Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego, San Diego, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - TORI - Oncology Care Med Assoc, San Gabriel, California
  - Kaiser Permanente Santa Teresa, San Jose, California
  - Kaiser Permanente San Rafael, San Rafael, California
  - Santa Barbara Hematology Oncology Medical Group, Santa Barbara, California
  - Santa Barbara II (Samsum Clinic) - TORI, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Santa Barbara Hematology/Oncology Medical Group, Inc, Solvang, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Olive View/UCLA Medical Center, Sylmar, California
  - Kaiser Permanente Medical Center Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Trivalley Oncology Hematology, Westlake Village, California
  - Westlake Infusion Center, Westlake Village, California
  - TORI - Oncology Care Med Assoc, Whittier, California
  - Medical Center of Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Center, Aurora, Colorado
  - Rocky Mountain Cancer Centers - Boulder, Boulder, Colorado
  - Penrose/St. Francis Healthcare System, Colorado Springs, Colorado
  - Rocky Mountain Cancer Center at the Pivillion- Fontanero, Colorado Springs, Colorado
  - Rocky Mountain Cancer Center - CO Springs, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla St. Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Center - Midtown, Denver, Colorado
  - Rocky Mountain Cancer Center - 9th Avenue, Denver, Colorado
  - Rocky Mountain Cancer Center - Rose, Denver, Colorado
  - University of Colorado, Denver, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Center, Lakewood, Colorado
  - Rocky Mountain Cancer Center - Dry Creek, Littleton, Colorado
  - Rocky Mountain Cancer Center- Sky Ridge, Lone Tree, Colorado
  - Rocky Mountain Cancer Center - Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Rocky Mountain Cancer Center, Parker, Colorado
  - Rocky Mountain Cancer Centers, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Washington Regional Cancer Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - SCRI - Florida Cancer Specialists- Bonita Springs, Bonita Springs, Florida
  - SCRI - Florida Cancer Specialists - Bradenton, Bradenton, Florida
  - Florida Cancer Specialists, Brandon, Florida
  - SCRI Florida Cancer Specialists - Cape Coral (1708), Cape Coral, Florida
  - SCRI Florida Cancer Specialists - Cape Coral (811), Cape Coral, Florida
  - Morton Plant Mease Health Care, Clearwater, Florida
  - SCRI Florida Cancer Specialists - Englewood, Englewood, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - SCRI Florida Cancer Specialists - Fort Myers (Hampshire), Fort Myers, Florida
  - SCRI Florida Cancer Specialists - Ft. Myers (Broadway), Fort Myers, Florida
  - SCRI Florida Cancer Specialists- Fort Myers (Veronica), Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Florida Cancer Institute - New Hope, Hudson, Florida
  - TORI-ICON - Shircl, Jacksonville, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Integrated Community Oncology Network (ICON), Jacksonville, Florida
  - TORI-ICON St.Aug, Jacksonville, Florida
  - CCOP, Jupiter Medical Cener, Jupiter, Florida
  - Ocala Oncology Center - Lady Lake, Lady Lake, Florida
  - Melbourne International Medicine Associates, Melbourne, Florida
  - Advanced Medical Specialties - AMS, Miami, Florida
  - Advanced Medical Specialists- Sunset, Miami, Florida
  - Advanced Medical Specialties - N Kendall (STE 300E), Miami, Florida
  - Advanced Medical Specialties - N. Kendall (STE 905E), Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - SCRI Florida Cancer Specialists - Naples (Goodlette), Naples, Florida
  - SCRI Florida Cancer Specialists - Naples (Pine), Naples, Florida
  - Florida Cancer Institute - New Hope, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - Tori-Icon, Orange Park, Florida
  - Florida Hospital, Orlando, Florida
  - Cancer Centers of Florida, P.A., Orlando, Florida
  - MD Anderson Cancer Center, Orlando, Florida
  - SCRI - Florida Cancer Specialists - Port Charlotte, Port Charlotte, Florida
  - Tori-Icon, Saint Augustine, Florida
  - SCRI Florida Cancer Specialists - Sarasota (Cattleman), Sarasota, Florida
  - SCRI- Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - SCRI - Florida Cancer Specialists - Armenia, Tampa, Florida
  - SCRI - Florida Cancer Specialists - Tampa, Tampa, Florida
  - SCRI Florida Cancer Specialists - Venice (Tamiami), Venice, Florida
  - SCRI Florida Cancer Specilaists - Venice, Venice, Florida
  - Cancer Centers of Florida, P.A., Winter Park, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Northwest Georgia Oncology Centers, Austell, Georgia
  - Northwest Georgia Oncology Centers, Carrollton, Georgia
  - Dublin Hematology/Oncology, Dublin, Georgia
  - Suburban Hematology-Oncology Associates, Lawrenceville, Georgia
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - SCRI Chattanooga Oncol & Hematol Assoc, PC - Ringgold, Ringgold, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Kaiser Permanente Hawaii - Moanalua Med Center, Honolulu, Hawaii
  - Cancer Care & Hematology Specialists of Chicagoland, Arlington, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - CCOP NorthShore University HealthSystem, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Edward Hospital, Naperville, Illinois
  - Cancer Care & Hematology Specialists of Chicagoland, Niles, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Carle Cancer Center, CCOP, Urbana, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland, Winfield, Illinois
  - Central Indiana Cancer Centers, Carmel, Indiana
  - Central Indiana Cancer Centers, Fishers, Indiana
  - Central Indiana Cancer Centers, Greenfield, Indiana
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Central Indiana Cancer Centers (E. County), Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Clarian Arnett Cancer Care, Lafayette, Indiana
  - Community Hospital, Munster, Indiana
  - Genesis Medical Center, Davenport, Iowa
  - Finley Hospital, Dubuque, Iowa
  - University of Iowa, Iowa City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Kansas Cty Cancer Center - West, Kansas City, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Kansas City Cancer Center (CBO), Overland Park, Kansas
  - Kansas CityCancer Centers - Southwest, Overland Park, Kansas
  - Kansas City Cancer Center, Shawnee Mission, Shawnee Mission, Kansas
  - SCRI Oncology Hematology Care, Inc. Crestview Hills (CVH), Crestview Hills, Kentucky
  - University of Kentucky Medical Center, Lexington, Kentucky
  - NortonHealtcare Inc., Louisville, Kentucky
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Christus St. Frances Cabrini Hospital, Alexandria, Louisiana
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Tulane University Medical Center, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Mercy Medical Center, Baltimore, Maryland
  - St. Joseph's Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - SCRI - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Chevy Chase Healthcare Management, LLC, Chevy Chase, Maryland
  - Maryland Oncology Hematology PA, Columbia, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Alliance Hematology Oncology PA, Owings Mills, Maryland
  - Penisula Regional Medical Center, Salisbury, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Alliance Hematology Oncology PA, Westminster, Maryland
  - Saint Anne's Hospital, Fall River, Massachusetts
  - Berkshire Hematology Oncology, P.C., Pittsfield, Massachusetts
  - CCOP, St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - CCOP - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - CCOP - St. John Hospital and Medical Center, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - CCOP - Genesys Regional Hospital, Flint, Michigan
  - CCOP - Hurley Medical Center, Flint, Michigan
  - McLaren Regional Medical Center, Flint, Michigan
  - CCOP - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ingham Regional Medical Center - Lansing, Lansing, Michigan
  - CCOP, Sparrow Health System, Lansing, Michigan
  - Lapeer Regional Hospital, Lapeer, Michigan
  - CCOP - St. Mary Mercy Hospital - Livonia, Livonia, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - Mount Clemens Regional Medical Center, Mount Clemens, Michigan
  - Memorial Healthcare, Owosso, Michigan
  - CCOP - St. Joseph Mercy Hospital - Oakland, Pontiac, Michigan
  - CCOP - St. Joseph Mercy Port Huron, Port Huron, Michigan
  - CCOP, William Beaumont Hospital, Royal Oak, Michigan
  - CCOP, St. Mary's Medical Center, Saginaw, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP, St. John Macomb Hospital, Warren, Michigan
  - Minnesota Oncology Hematology-Burnsville, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - St. Luke's Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Minnesota Oncology Hematology-Edina, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA - Maplewood, Maplewood, Minnesota
  - St. John's Hospital Northeast/HealthEast, Inc., Maplewood, Minnesota
  - Minnesota Oncology Hematology-Minneapolis, Minneapolis, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - North Memorial Health Care, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - Minnesota Hematology Oncology-St. Paul, Saint Paul, Minnesota
  - Minnesota Oncology Hematology, Woodbury, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - University of Missouri-Ellis Fischel, Columbia, Missouri
  - Kansas City Cancer Center - Central, Kansas City, Missouri
  - Saint Luke's Hospital, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Kansas City Cancer Center - South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Kansas City Cancer Center - North, Kansas City, Missouri
  - Kansas City Cancer Centers - East, Lee's Summit, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - St. Elizabeth Community Health Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - CCOP, Missouri Valley Cance Consortium, Omaha, Nebraska
  - Creighton University Cancer Center, Omaha, Nebraska
  - Alegent Health Midlands Hospital, Papillion, Nebraska
  - Comprehensive Cancer Centers of Nevada (Siena), Henderson, Nevada
  - US Oncology West Region Office (Horizon Ridge), Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada (Wigwam), Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada (Peak Dr.), Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada (Southern Hills), Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada (Twain), Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Hematology-Oncology Associates of NNJ, PA, Morristown, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Clare's Center at Parsippany Commons, Parsippany, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Sparta Cancer Center, Sparta, New Jersey
  - Texas Oncology PA Las Cruces, Las Cruces, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - New York Oncology Hematology PC-Albany, Albany, New York
  - New York Oncology Hematology, PC at Albany Medical Center, Albany, New York
  - Amsterdam Community Cancer Program, Amsterdam, New York
  - Interlakes Oncology Hematology PC, Brockport, New York
  - Interlakes Oncology & Hematology, P.C., Canandaigua, New York
  - Interlakes Oncology Hematology PC, Geneva, New York
  - Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - New York Oncology Hematology, P.C. at Cavell Cancer Treatment Program, Hudson, New York
  - New York Oncology Hematology, PC, Latham, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - CCOP, Long Island Jewish Medical Center, New Hyde Park, New York
  - New York University School of Medicine, New York, New York
  - New York Oncology Hematology PC, Rexford, New York
  - Interlakes Oncology Hematology PC - White Spruce, Rochester, New York
  - Interlakes Oncology Hematology PC- Long Pond, Rochester, New York
  - University Hospital and Medical Center - SUNY Stony Brook, Stony Brook, New York
  - Troy Cancer Treatment Program, Troy, New York
  - Alamance Regional Medical Center, Burlington, North Carolina
  - Cancer Centers of North Carolina, Cary, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - CCOP Carolinas HealthCare System, Charlotte, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - Regional Cancer Care, PA, Durham, North Carolina
  - Virginia Oncology Associates, Elizabeth City, North Carolina
  - Cape Fear Valley Medical Center Cancer Center, Fayetteville, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - CCOP, Moses Cone Health System-Regional CA Cntr, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Margaret R. Pardee Memorial Hospital, Hendersonville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Cancer Centers of North Carolina, Raleigh, North Carolina
  - Cancer Centers of North Carolina- North Raleigh, Raleigh, North Carolina
  - CCOP Forsyth Memorial Hospital, Winston-Salem, North Carolina
  - Innovis Health, Fargo, North Dakota
  - Akron City Hospital, Akron, Ohio
  - Aultman Hospital, Canton, Ohio
  - SCRI Oncology Hematology Care, Inc. - Cincinnati (TFT), Cincinnati, Ohio
  - SCRI Oncology Hematology Care, Inc - Cincinnati (AND), Cincinnati, Ohio
  - SCRI Oncology Hematology Care, Inc. - Cincinnati (KWD), Cincinnati, Ohio
  - SCRI Oncology Hematlogy Care, Inc. - Cincinnati (RPR), Cincinnati, Ohio
  - SCRI Oncology Hematology Care, Inc - Cincinnati (BAM), Cincinnati, Ohio
  - SCRI Oncology Hematology Care, Inc. Cincinnati (WST), Cincinnati, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - HemOnc Care, Inc., Fairfield, Ohio
  - Atrium Medical Center - Middletown Regional Hosp, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - SCRI Oncology Hematology Care, Inc. - Hamilton (HAM), Hamilton, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - SCRI Oncology Hematology Care, Inc. - Wilmington (WLM), Wilmington, Ohio
  - St. Charles Medical Center - Bend, Bend, Oregon
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Northwest Cancer Specialists-Portland, Portland, Oregon
  - Providence Medical Center, Portland, Oregon
  - Northwest Cancer Specialists- St. Vincent, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Northwest Cancer Specialists- Rose Qtr, Portland, Oregon
  - Williamette Valley Cancer Institute and Research Center, Springfield, Oregon
  - Celilo Center for Cancer Care, The Dalles, Oregon
  - Northwest Cancer Specialists-Tualatin, Tualatin, Oregon
  - Geisinger Clinic, Danville, Pennsylvania
  - Oncology Hematology Associates of Northern PA, DuBois, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Community Hopital, Ephrata, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Medical Oncology Associates, Kingston, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Rittenhouse Hematology/Oncology, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Albert Einstein Healthcare Network, Philadelphia, Pennsylvania
  - Allegheny General Hospital/Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Hematology and Oncology Associates of NEPA, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Associates in Hematology-Oncology, PC at Crozer Regional Cancer Center, Upland, Pennsylvania
  - Reading Hospital and Medical Center, West Reading, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Roper Hosp & Med Asso (Care Alliance Health), Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - SCRI - South Carolina Oncology Associates - Stoneridge, Columbia, South Carolina
  - Cancer Centers of the Carolinas Easley, SC, Easley, South Carolina
  - Georgetown Hospital System, Georgetown, South Carolina
  - Cancer Centers of the Carolinas (Butternut), Greenville, South Carolina
  - Cancer Centers of the Carolinas-W. Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas (International), Greenville, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Spartanburg Regional Healthcare System, Spartanburg, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Avera McKenna Hospital, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - CCOP, Sanford Cancer Center - Oncology Clinic, Sioux Falls, South Dakota
  - SCRI Chattanooga Oncol & Hematol Assoc, PC - Chattanooga, Chattanooga, Tennessee
  - SCRI Tennessee Oncology - PLLC Franklin, Franklin, Tennessee
  - SCRI Tennessee Oncology- Gallatin, Gallatin, Tennessee
  - SCRI Tennessee Oncology, PLLC Hermitage, Hermitage, Tennessee
  - SCRI Chattanooga Oncol & Hematol Assoc, PC Hixson, Hixson, Tennessee
  - CCOP Holston Valley Medical Center, Kingsport, Tennessee
  - SCRI Tennessee Oncology Lebanon, Lebanon, Tennessee
  - SCRI Tennessee Oncology Murfreesboro, Murfreesboro, Tennessee
  - SCRI - Tennessee Oncology PLLC, Nashville, Tennessee
  - SCRI Tennessee Oncology, PLLC (Harding), Nashville, Tennessee
  - SCRI Tennessee Onclogy, PLLC (Dickerson), Nashville, Tennessee
  - SCRI Tennessee Oncology, PLLC (Wallace), Nashville, Tennessee
  - Tennessee Oncology, Shelbyville, Tennessee
  - SCRI Tennessee Oncology, PLLC Smyrna, Smyrna, Tennessee
  - Texas Cancer Center - Abilene South, Abilene, Texas
  - Texas Oncology PA - Amarillo, Amarillo, Texas
  - Texas Oncology PA - Arlington North, Arlington, Texas
  - Texas Onclogy - Arlington South, Arlington, Texas
  - Texas Oncology Central Austin, Austin, Texas
  - Texas Oncology Cancer Center - Balcones, Austin, Texas
  - South Austin Cancer Center, Austin, Texas
  - Southwest Regional Cancer Center- North, Austin, Texas
  - Texas Oncology North Austin- Renfert, Austin, Texas
  - Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Edwards Cancer Center - Bedford, Bedford, Texas
  - Texas Oncology PA - Harris HEB, Bedford, Texas
  - Texas Oncology, PA - Cedar Park, Cedar Park, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Oncology PA- Presbyterian, Dallas, Texas
  - Methodist Charlton Cancer Center, Dallas, Texas
  - Texas Oncology- Sammons CC, Dallas, Texas
  - Texas Cancer Center, Denton, Texas
  - El Paso Cancer Treatment Center - West, El Paso, Texas
  - El Paso Cancer Treatment Center - East, El Paso, Texas
  - Texas Oncology - 8th Avenue, Fort Worth, Texas
  - Texas Oncology at Klabzuba, Fort Worth, Texas
  - Texas Oncology PA - 12th Avenue, Fort Worth, Texas
  - Southwest Fort Worth Cancer Center, Fort Worth, Texas
  - San Antonio Tumor and Blood Clinic, Fredericksburg, Texas
  - Texas Oncology PA, Garland, Texas
  - Texas Oncology, Grapevine, Texas
  - Texas Oncology PA - Frostwood, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - San Antonio Tumor and Blood Clinic, Kerrville, Texas
  - Lake Vista Cancer Center, Lewisville, Texas
  - Longview Cancer Center, Longview, Texas
  - Joe Arrington Cancer Research & Treatment Center, Lubbock, Texas
  - South Texas Cancer Center - McAllen, McAllen, Texas
  - Texas Cancer Center of Mesquite, Mesquite, Texas
  - Allison Cancer Center, Midland, Texas
  - HOAST - New Braunfels, New Braunfels, Texas
  - Texas Oncology - Odessa, Odessa, Texas
  - Paris Regional Cancer Center, Paris, Texas
  - North Texas Regional Cancer Center, Plano, Texas
  - Texas Oncology Plano West Cancer Center, Plano, Texas
  - Texas Oncology Seton Williamson, Round Rock, Texas
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - Cancer Care Centers of South Texas- Brooklyn, San Antonio, Texas
  - Cancer Care Centers of South Texas - Loop 410, San Antonio, Texas
  - HOAST - Medical Drive, San Antonio, Texas
  - San Antonio Tumor and Blood Clinic - M.Oak, San Antonio, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Texas Oncology - San Marcos, San Marcos, Texas
  - Texas Cancer Center, Sherman, Texas
  - Texas Oncology Cancer Center - Sugar Land, Sugar Land, Texas
  - US Oncology, The Woodlands, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology Cancer Care and Research Center, Waco, Texas
  - Texas Oncology - Clear Lake, Webster, Texas
  - South Texas Cancer Clinic, Weslaco, Texas
  - Texoma Cancer Center, Wichita Falls, Texas
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Huntsman Cancer Inst. at the University of Utah- Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Southwestern Regional Cancer Center (SWORD), Bennington, Vermont
  - Arlington Fairfax Hematology Oncology, Arlington, Virginia
  - Virginia Oncology Associates - Medical Pkwy, Chesapeake, Virginia
  - Oncology and Hematology Associates of SW VA, Inc, Christiansburg, Virginia
  - Fairfax Northern VA Hematology-Oncology PC, Fairfax, Virginia
  - Fair Oaks Office, Fairfax, Virginia
  - Fairfax-Northern Virginia Hematology-Oncology PC, Gainesville, Virginia
  - Virginia Oncology Associates, Hampton, Virginia
  - Fairfax-Northern Virginia Hematology-Oncology PC, Leesburg, Virginia
  - SCRI Virginia Cancer Institute (Flank), Mechanicsville, Virginia
  - SCRI Virginia Cancer Institute, Midlothian, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates - Lake Wright, Norfolk, Virginia
  - SCRI Virginia Cancer Institute (6605), Richmond, Virginia
  - SCRI Virginia Cancer Institute (1401), Richmond, Virginia
  - MBCCOP, Virginia Commonwealth University, Richmond, Virginia
  - Oncology and Hematology Associates of SW VA, Inc, Roanoke, Virginia
  - Oncology and Hematology Associates of SW VA, Inc, Salem, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
  - Virginia Oncology Associates, Williamsburg, Virginia
  - Fairfax Northern Virginia Hematology-Oncology - Winchester, Winchester, Virginia
  - Fairfax-Northern Virginia Hematology-Oncology PC, Woodbridge, Virginia
  - Oncology and Hematology Associates of SW VA, Inc, Wytheville, Virginia
  - Highline Medical Oncology, Burien, Washington
  - Puget Sound Cancer Center- Edmonds, Edmonds, Washington
  - Columbia Basin Hematology and Oncology, Kennewick, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Puget Sound Cancer Center - Seattle, Seattle, Washington
  - Cancer Care Northwest-South, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Cancer Care Northwest-Radiation Therapy (XRT), Spokane, Washington
  - Cancer Care Northwest- Valley - Mission, Spokane, Washington
  - Cancer Care Northwest-North - Holland, Spokane, Washington
  - Evergreen Hematology & Oncology (Farwell), Spokane, Washington
  - Northwest Cancer Specialists-136th Ave, Vancouver, Washington
  - Northwest Cancer Specialists-134th St., Vancouver, Washington
  - Yakima Valley Memorial Hospital - North Star Lodge, Yakima, Washington
  - Raleigh Regional Cancer Center, Beckley, West Virginia
  - CAMC Health Education & Research Institute, Inc., Charleston, West Virginia
  - West Virginia University Hospitals Inc., Morgantown, West Virginia
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Wheeling Hospital, Wheeling, West Virginia
  - Marshfield Clinic Chippewa Falls Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Regional CA Cntr - Sacred Heart Hospital, Eau Claire, Wisconsin
  - CCOP, St. Vincent Hospital, Green Bay, Wisconsin
  - CCOP, St. Mary's Hospital Medical Center, Green Bay, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Froedtert Hospital, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic Minocqua Center, Minocqua, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic Rice Lake Center, Rice Lake, Wisconsin
  - Marshfield Clinic Cancer Care at St. Michael's Hospital, Stevens Point, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Women's Pavilion of Aurora West Allis Medical Center, West Allis, Wisconsin
  - CCOP Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
- Ireland (11):
  - Bon Secours Hospital, Cork, CK
  - Letterkenny General Hospital, Letterkenny, DL
  - Mater Private Hospital, Dublin, DN
  - Beaumont Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - Mater Misericordiae, Dublin
  - St James' Hospital, Dublin
  - St. James' Hospital, Dublin
  - University College Hospital, Galway
  - Sligo General Hospital, Sligo
  - Waterford Regional Hospital, Waterford

REFERENCES:
- [Derived] Geyer CE Jr, Blum JL, Yothers G, Asmar L, Flynn PJ, Robert NJ, Hopkins JO, O'Shaughnessy JA, Rastogi P, Puhalla SL, Hilton CJ, Dang CT, Gomez HL, Vukelja SJ, Lyss AP, Paul D, Brufsky AM, Colangelo LH, Swain SM, Mamounas EP, Wolmark N. Long-Term Follow-Up of the Anthracyclines in Early Breast Cancer Trials (USOR 06-090, NSABP B-46-I/USOR 07132, and NSABP B-49 [NRG Oncology]). J Clin Oncol. 2024 Apr 20;42(12):1344-1349. doi: 10.1200/JCO.23.01428. Epub 2024 Feb 9. PMID 38335467